CLINICAL TRIAL: NCT06726122
Title: Clinical Study to Evaluate the Efficacy and Safety of Matrix Pro Treatment for Facial, Submental and Neck Laxity
Brief Title: Clinical Study to Evaluate the Efficacy and Safety of Matrix Pro Treatment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFX22003_EU
Record Dates: First submitted 2024-12-03; First posted 2024-12-10 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Skin Laxity; Wrinkle; Skin Condition
MeSH Terms: conditions — Cutis Laxa; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Matrix Pro Treatment Group (Experimental): Study subjects receive up to three (3) study treatments with the Matrix Pro applicator
  Interventions: Device: Profound Matrix

INTERVENTIONS:
Device: Profound Matrix — Treatment visits are limited to up to three (3) study treatments (with treatment intervals 6 weeks ± 2 weeks).

SUMMARY:
This is a non-randomized, multi-center, open-label, prospective clinical trial evaluating clinical treatments with the Matrix Pro Applicator for the improvement of facial and/or submental and neck laxity.

DETAILED DESCRIPTION:
Eligible participants will receive up to three treatments with the Matrix Pro Applicator of the Profound Matrix System to address facial and neck laxity. Treatments will be approximately 6 weeks apart (± 2 weeks). All participants will undergo follow-up evaluations at 1 month (4 weeks ± 2 weeks) and 3 months (13 weeks ± 2 weeks) after the final treatment. Additional follow-up visits may be required per Sponsor and PI discretion

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between 18 to 84 years of age with Fitzpatrick Skin Type I - VI.
2. Willing to receive Profound Matrix treatments with Matrix Pro applicator
3. Able and willing to comply with the treatment/follow-up schedule and comply with all study (protocol) requirements.
4. Willing to provide signed, informed consent to participate in the study
5. Willing to have photographs and images taken of the treated areas to be used in evaluations, publications, presentations, and marketing materials (Subject identity will be masked).

Exclusion Criteria:

Any of the following will exclude the subject from the study:

1. Pregnant or planning to become pregnant, having given birth less than 3 months prior to enrollment into the study, and/or breast feeding
2. Pacemaker or internal defibrillator or any active electrical implant anywhere in the body
3. Superficial metal or other implants in the treatment area, except superficial dental implants, unless the implants can be removed or covered with rolled gauze during treatment
4. Skin cancer in the treatment area or history of melanoma
5. History of current cancer and/or subject has undergone chemotherapy within the last 12 months
6. Severe concurrent conditions, such as cardiac disorders
7. Impaired immune system or use of immunosuppressive medications, except for topical products and inhaler medications per investigator discretion
8. Herpes Simplex Virus (HSV) in the intended treatment area unless treated following a prophylactic regimen
9. Poorly controlled endocrine disorders such as poorly controlled diabetes
10. Active skin condition in the treatment area such as skin infection, sores, psoriasis, eczema, rash, or open wounds
11. History of abnormal wound healing, keloid, or hypertrophic scar formation, as well as very thin or fragile skin
12. History of collagen vascular disease or vasculitic disorders
13. Known allergy to medication to be used during treatments such as allergy to topical anesthetic (e.g., lidocaine)
14. History of systemic corticosteroid therapy in past six months
15. Tattoos or permanent makeup in the intended treatment area
16. Excessively tanned skin
17. Facelift in the last 12 months
18. Aesthetics treatments/procedures (e.g., facial resurfacing and deep chemical peeling) within the last 4 months within the intended treatment area
19. Neuromodulator injections (e.g., Botox®), collagen, non-permanent dermal filler, fat injections or other methods of augmentation with injected biomaterial in the intended treatment area within the last 3 months
20. Permanent synthetic fillers (e.g., silicone) in the intended treatment area
21. Absorbable facial threads within the last 12 months or non-absorbable facial threads within the intended treatment area
22. In the opinion of the Investigator, the subject is unwilling or unable to adhere to the study requirements or is otherwise unsuitable for study participation

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of change in facial, submentum, and neck laxity | From subject enrollment to completion of 3-month follow-up visit, up to 32 weeks.
  Evaluation of change in facial, submentum, and neck laxity based on correct identification of subject's post-treatment photograph by at least 2 of the 3 independent blinded reviewers.

CONTACTS AND LOCATIONS:
Overall Officials: Konika Schallen, MD, Study Director — Candela Corporation
Locations (3):
- Kliniek voor Esthetische Geneeskunde, Amsterdam, EK, Netherlands
- United Kingdom (2):
  - Illuminate Skin & Wellness Clinic, Kings Hill, Kent
  - GHB Clinic, London

IPD SHARING:
Plan to Share IPD: No